CLINICAL TRIAL: NCT04095429
Title: Expect Respect Middle School: Preventing Serious and Lethal Violence Among Youth With Prior Violence Exposure
Brief Title: Expect Respect Middle School Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Elizabeth Miller, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY18080006; R01CE002981 (NIH)
Record Dates: First submitted 2019-09-06; First posted 2019-09-19 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Adolescent Behavior; Violence in Adolescence; Group, Peer; Violence, Non-accidental; Violence, Sexual; Violence, Physical; Violence, Domestic; Emotional Abuse; Coping Skills; Communication, Personal
MeSH Terms: conditions — Adolescent Behavior; Coitus; Communication

STUDY DESIGN:
Intervention Model Description: This cluster-randomized school-based study will examine the effectiveness of a support group-based teen dating violence (TDV) and sexual violence (SV) prevention program on the primary prevention of serious (and potentially lethal) violence perpetration among middle school students (both male and female-identified) already exposed to violence. The study will be located in western Pennsylvania across 36 middle schools (anticipated number of 'clusters'), randomized either to receive the "Expect Respect" program (i.e., intervention schools, n=18) or to an enhanced usual care condition (n=18 schools).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Expect Respect Support Group (Experimental): Experimental: Expect Respect Support Group Expect Respect is a program intended to create safe, trauma-informed space for young people who have been exposed to violence, to promote positive bystander intervention and healthy relationship skills, to alter norms that foster TDV/SV perpetration, and reduce violence perpetration through weekly support groups with students at elevated risk for such perpetration. Youth with prior history of exposure to violence are invited to in-school gender specific support groups that take place over 24 in-classroom sessions.
  Expect Respect addresses violence perpetration prevention with youth already exposed to violence by recognizing violence as a problem that is fueled by gender norms that promote dominance and challenging the need to control and exert power in relationships especially with the use of violence, while simultaneously strengthening emotion regulation, social skills, and connectedness.
  Interventions: Behavioral: Expect Respect
- Enhanced Usual Care (Active Comparator): Comparator: Enhanced Usual Care The control arm will receive enhanced usual care. Enhanced care means that the investigators will ensure each school has information, resource lists, and connection to services for individual youth who are referred to the study, including warm referrals to victim service agencies, behavioral health services, as well as resources (e.g., assistance with food insecurity, and so forth).
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: Expect Respect — Expect Respect is a 24 session curriculum designed to support middle school students to increase skills in emotion regulation, relationship skills, communication, and positive bystander intervention behaviors.
  Arms: Expect Respect Support Group
Behavioral: Enhanced Usual Care — Participants will be connected via a warm referral to available individual behavioral health supports and resources in their community that can support them.
  Arms: Enhanced Usual Care

SUMMARY:
This cluster-randomized school-based study will examine the effectiveness of a teen dating violence (TDV) and sexual violence (SV) prevention program called Expect Respect for preventing serious violence perpetration among middle school students.

DETAILED DESCRIPTION:
This cluster-randomized controlled school-based study will examine the effectiveness of a support group-based teen dating violence (TDV) and sexual violence (SV) prevention program on the primary prevention of serious (and potentially lethal) violence perpetration among middle school students (both male and female-identified) who have prior exposure to trauma and violence. Expect Respect gender-specific support groups are for youth with prior history of exposure to violence including witnessing domestic violence, loss of loved one to homicide, TDV, and SV.

Expect Respect is a theory and research-informed program intended to alter norms condoning violence and rigid gender expectations that foster violence perpetration, promote bystander intervention, and reduce TDV/SV perpetration. Implemented by trained facilitators, the 24-session curriculum focuses on gender equity and respect, recognizing abuse and impact on self and others, regulating emotions, skills for healthy relationships, and becoming active proponents of safe and healthy relationships.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be in grades 7-8
* Participants must be referred by school personnel
* Participants must speak English

Exclusion Criteria:

* Not in 7th- 8th grade
* Not referred to the group by school personnel
* Does not speak English

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Participants will be placed in gender-specific support groups based on how they identify their gender.
Enrollment: 635 (Actual)
Dates: Start 2019-10-03 (Actual); Primary Completion 2021-08-17 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in self-reported recent (past 3 months) violence perpetration at End of Program | End of program (average 24-30 weeks after baseline, Time 2 - primary endpoint)
  Summary score of violence perpetration likely to result in serious injury or death (physical and sexual TDV - 4 items, SV - 5 items, threats with a weapon - 1 item, and physical fighting - 1 item), calculated as one point for each behavior endorsed and then summed (possible range: 0-11).
Change from baseline in self-reported recent (past 3 months) violence perpetration at one year after baseline | One year after baseline (Time 3)
  Summary score of violence perpetration likely to result in serious injury or death (physical and sexual TDV - 4 items, SV - 5 items, threats with a weapon - 1 item, and physical fighting - 1 item), calculated as one point for each behavior endorsed and then summed (possible range: 0-11).

SECONDARY OUTCOMES:
Change from baseline in frequency of weapon carrying at End of Program | End of program (average 24-30 weeks after baseline, Time 2 - primary endpoint)
  Number of times carrying a weapon in past 30 days (self-reported)
Change from baseline in frequency of weapon carrying at one year after baseline | One year after baseline (Time 3)
  Number of times carrying a weapon in past 30 days (self-reported)
Change from baseline in positive bystander behaviors at End of Program | End of program (average 24-30 weeks after baseline, Time 2 - primary endpoint)
  Past 3 month positive bystander behavior in participants when witnessing disrespectful and harmful behavior among peers comparing baseline and follow up summary scores. Participants report if they have witnessed each of 9 peers' abusive behaviors in the past 3 months and if witnessed, how they responded (whether they intervened to interrupt the behavior, provided support to the person being harmed). One point is given for reporting at least 1 positive intervention for each abusive behavior witnessed; points are added to create a summary score (possible range: 0-9).
Change from baseline in positive bystander behaviors at one year after baseline | One year after baseline (Time 3)
  Past 3 month positive bystander behavior in participants when witnessing disrespectful and harmful behavior among peers comparing baseline and follow up summary scores. Participants report if they have witnessed each of 9 peers' abusive behaviors in the past 3 months and if witnessed, how they responded (whether they intervened to interrupt the behavior, provided support to the person being harmed). One point is given for reporting at least 1 positive intervention for each abusive behavior witnessed; points are added to create a summary score (possible range: 0-9).

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Miller, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The research team anticipates making deidentified data from this study available to other researchers 12 months after study completion.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 12 months after study completion; indefinitely
Access Criteria: Researchers must contact the PI (Miller) with any requests for use of the data.